CLINICAL TRIAL: NCT04886024
Title: The Serum Ages Levels in Patients With Endometriosis
Brief Title: Evaluation of Serum Ages Levels in Patients With Endometriosis
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: endo-serum ages levels
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Endometriosis
Keywords: AGES (Advanced Glycation End Products)
MeSH Terms: conditions — Endometriosis | interventions — Glycation End Products, Advanced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women with endometriosis: It consists of women between the ages of 18-45 who have been diagnosed with endometriosis by surgery or ultrasonography.
  Interventions: Other: Advanced Glycation End Products (AGEs)
- control: It consists of healthy women between the ages of 18-45
  Interventions: Other: Advanced Glycation End Products (AGEs)

INTERVENTIONS:
Other: Advanced Glycation End Products (AGEs) — Advanced Glycation End Products (AGEs) releated with energy metabolism, In this study, the possible relationship between the serum levels of Advanced Glycation End Products (AGEs) of endometriosis patients and the disease and its stage is evaluated.

SUMMARY:
Serum AGES (Advanced Glycation End Products) levels of endometriosis patients are compared with a group of healthy volunteers of the same age.

DETAILED DESCRIPTION:
Serum AGES (Advanced Glycation End Products) levels are compared with 45 endometriosis patients and 45 healthy volunteers of the same age. The energy metabolism of the endometriosis group and its possible relationship with the endometriosis stage will be compared since AGES (Advanced Glycation End Products) gives information about the energy metabolism of the people.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with endometriosis (Surgery or ultrasound)
* Women without endometriosis

Exclusion Criteria:

* Women without endometriosis women who are only suspected endometriosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women aged 18-45 diagnosed with endometriosis (surgery or ultrasound)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Serum Advanced Glycation End Products (AGEs) levels in women with endometriosis | 8 months
  Serum Serum Advanced Glycation End Products (AGEs) levels involved in inflammation and energy metabolism are compared between endometriosis and healthy control group

SECONDARY OUTCOMES:
Comparison of the relationship between serum Serum Advanced Glycation End Products (AGEs) level and endometriosis stage | 8 months
  By comparing the relation of serum Advanced Glycation End Products (AGEs) level with the stage of endometriosis, its relation with serum level in patients with advanced and early stage endometriosis will be examined. The possible effect of Advanced Glycation End Products (AGEs) on disease pathogenesis will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided